CLINICAL TRIAL: NCT04598971
Title: Consequences of UTI on Urine pH
Brief Title: Urine pH and Urinary Tract Infection
Acronym: PHURINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Olivier Bonny, Associate professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2020-00779
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Urinary Tract Infections; Urinary Stone
Keywords: urine pH
MeSH Terms: conditions — Urinary Tract Infections; Urinary Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystitis: Patients with lower UTI will be included in this group
- Pyelonephritis: Patients with higher UTI will be included in this group

SUMMARY:
Urinary tract infections (UTI) affect the urine pH and may lead to salt precipitation such as struvite. Bacteria with urease activity are known to alkalinise urine, but not much is known on how pH is changing over time during UTI.

This study aims at following urine pH progression at the time of diagnosis of UTI and during the treatment phase.

Description of the change in urine pH over time will help understanding the risk of struvite formation and potential timing of intervention.

DETAILED DESCRIPTION:
Adults presenting with UTI symptoms will be screened for infection and instructed to monitor urine pH during the course of treatment and 1 week after. Urine pH will be measured by the patients using calibrated pH-stix. Type of bacteria, antibiotics, and the type of diet will be monitored during the study.

ELIGIBILITY:
Group 1. Cystitis

Inclusion Criteria:

* Symptoms of dysuria, pollakiuria, no fever AND
* urine-stix positive for leucocytes OR positive culture (>10E5 cfu/ml)

Group 2. Pyelonephritis

Inclusion Criteria:

* Unilateral flank pain, pollakiuria, dysuria, fever (>38.5°C) AND
* urine-stix positive for leucocytes OR positive culture (>10E5 cfu/ml)

Exclusion Criteria (both groups):

* known urinary tract anatomic abnormalities
* Presence of a urine catheter
* Sepsis - septic shock
* Patient taking drug interfering with urine pH (diuretics, citrate, acetazolamide, topiramate,...)
* Patients with UTI diagnosed in the preceding month
* Patients having received antibiotics during the preceding month
* Male patient with a diagnosis of prostatitis
* Presence of infected kidney cyst
* Patient with diabetes
* Pregnant female
* Patient with obstructive pyelonephritis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient consulting the primary care unit of the medical outpatient clinic UniSanté in Lausanne will be asked to participate.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
Urine pH | 21 days
  Urine pH is monitored by the patient every morning during the treatment phase and 7 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bonny, MD-PhD, Principal Investigator — CHUV-Lausanne
Locations (1):
- UniSanté, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No